CLINICAL TRIAL: NCT05587777
Title: REsearch on BrEast Cancer Induced Chronic Conditions Supported by Causal Analysis of Multi-source Data
Brief Title: Monitoring of Chronic Conditions in Breast Cancer
Acronym: REBECCA-1
Status: Recruiting | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1234
Record Dates: First submitted 2022-09-26; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer; Chronic Fatigue Syndrome
Keywords: fatigue; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue Syndrome, Chronic; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — microRNA, circulating tumor DNA, metylation of DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild Cancer Related Fatigue: After treatment(6 months from inclusion) is ended a fVAS < 50
- Cancer related Fatigue: After treatment (6 months from inclusion) with fVAS ≥ 50 mm or a rise of fVAS of ≥ 25 mm.
- Healthy control: Healthy women matches with age
  1. 50-70: women attending the mammography screening
  2. 19-50: invitation in newspaper, flyers and posters

SUMMARY:
REBECCA-1 is an observational study. Clinical research is undergoing a revolutionary change. The use of electronic patient records (EHR), digital registers, smartphones etc will create "real-world data" (RWD) that provides great opportunities for advancing clinical research, but so far this opportunity has been little exploited. The REBECCA -1 study will observe and monitor fatigue in breast cancer survivors. Investigators will use self reported questionnaires (PROM-data), blood tests and objective regulations like the REBECCCA -1 smart watch that will register amount of steps every day, leaving the house, visiting friends, cafes etc. There will be three observational arms; 1.high fatigue, 2. low fatigue and 3. a healthy control arm. After the patients have finished their treatment, they will receive the REBECCA smart watch, a REBECCA app on the smart phone and a REBECCA plus device on their computer, The next offend are also invited to report their evaluation through the same apps. The observational time will be 1 year and comparison between the subjective PROM data , the objective REBECCA watch and the biological samples will be obtained.

DETAILED DESCRIPTION:
Detailed Description:

1. Background:

   Clinical research is undergoing revolutionary changes by use of electronic patient records (EHR), digital registers and smartphones. The widespread use of portable devices have led to possibilities to collect "real-world data" (RWD) that provides great opportunities for advancing clinical research.

   Fatigue or exhaustion is one of the most common and most annoying late side effects after breast cancer treatment. Cancer Related Fatigue (CRF) may be elevated even before starting treatment and generally increases in intensity during treatment . It can also persist for years after completion of treatment in otherwise healthy cancer survivors and studies suggest that up to a third experience persistent fatigue for up to 10 years after being diagnosed with cancer. CRF is multi-dimensional and can have physical, mental and emotional manifestations, including general weakness, decreased concentration or attention, decreased motivation or interest in participating in regular activities, as well as emotional lability. Fatigue has also been shown to have a negative impact on work, social relationships, mood and daily activities and causes a significant reduction in overall quality of life during and after treatment for the patients affected. Thus, studying of RWD in CRF will be an appropriate method and design. As far as known this has not been done before.

   The biological mechanisms associated with the development of CRF may involve inflammatory processes contribute to fatigue during and especially after cancer treatment. Various cytokines may be produced during cancer treatment in response to tissue damage from radiation or chemotherapy. Inflammatory candidate biomarkers include Interleukin (IL) 1b, IL6, IL10, IL-17, IL1βRa and IL1-RII 32, 33. Heat shock Protein (HSP) 90 is another current biomarker candidate as it has been shown to reflect the severity of fatigue in patients with Crohn's disease.
2. Rationale behind the REBECCA project

   By using multi-source RWD in clinical studies, it will be possible to monitor the quality of life of patients and have a unique opportunity to map the challenges patients have in their daily lives in terms of work life participation, physical activity, social activity / relationships and their concerns. At the same time, the investigators will explore whether different immunological candidate biomarkers can provide prognostic information related to the development of fatigue in this patient group.
3. Objectives

   REBECCA-1 is an observational study in which a REBECCA smartwatch will be used to monitor the quality of life and fatigue in breast cancer patients
4. Spesific aims include:

   * Evaluating whether the use of REBECCA-collected patient information (i.e. collection of continuous RWDs and PROMs) will provide better insight into fatigue in breast cancer survivors.
   * Evaluating immunological biomarkers such as HSP90, IL1b, IL6, IL10, IL-17, IL1βRa, IL1-RII, HPX, CFB, APOA4 and Serpin-F1 and DNA methylation patterns.
5. Study design

   The REBECCA-1 sub-study: Characterize the quality of life and late effects in breast cancer patients.

   In REBECCA-1, participants will be included in 3 groups à n = 49 Two of the groups include breast cancer patients. After treatment, the patient will be assigned to one of the two study arms as described below. The third arm is a control group consisting of healthy women between 19 and 70 years.

   After undergoing treatment (surgery, chemotherapy given neoadjuvant or adjuvant and radiation), the breast cancer patients will again fill in PROM data and submit biological material and be assigned to the "CRF arm" and "Mild CRF arm", respectively.

   "Cancer Related Fatigue (CRF) arm" n = 49: The participants who after evaluation of the form VAS-fatigue have a change of f-VAS> 25mm from the time of inclusion to evaluation after completion of treatment and / or fVAS score> = 50 mm are stratified into the group "CRF arm".

   "Mild Cancer Related Fatigue (mild CRF) arm" n = 49: Patients with a final fVAS score <50mm is randomized to the group "Mild CRF arm".

   All participants will be able to borrow a smartwatch during the observation period, which they must wear for 12 months (i.e. from month 6 to month 18). In addition, the participants must install a REBECCA patient app on their mobile and a plug-in on their PC in order to obtain objective RWD related to the participants' quality of life and lifestyle over the next 12 months. The data collected by means of these devices is described in the figure which shows which data is collected via the smartwatch and the mobile phone

   At all time points i.e. at diagnosis, 6, 12 and 18 months after the time of inclusion, patient reported outcome measures (PROMs), medicine list, biological samples and RWD from the smart watch system on REBECCA platform from all the participants in all three subgroups.
6. REAL WORLD DATA COLLECTION

   A. Smartwatch:

   Acceleration, pulse, Activity sessions (type of exercise (running, walking, walking, cycling Length of activity(minutes, training distance (km) and altitude meters Intensity level(number of calories, intensity B. Smartphone and mobile apps
   * GPS positions (movement pattern)
   * Answer to questionnaires
   * Photo initiated in the Rebecca app (related to meals/eating habits and environment)
   * Publicity available data from map services location and environmental. C. REBECCA. PC plug in internet from *Social media such as Facebook, You Tube etc., D. REBECCA companion app (optional) *answer questions about the patient's quality of life , symptoms and environment
7. Patient Reported Outcome Measures (PROMs)

   Patient-reported data (PROMs) related to lifestyle, quality of life, working conditions, sleep and medication use will also be collected in REBECCA. For this purpose, the investigators will both use standardized PROM forms (ΕORTC-QLQ-BR2340, SF-3641, ΕORTC-QLQ-C3042, HAD43, FSS44, FQ45 og VAS-fatigue34, 46, 47) and self-report form.
8. Collection and analyses of blod-, urine- and faeces samples

   All patients included in the REBECCA-1 sub-study will be asked to give blood, urine and faeces samples i.) at the time of diagnosis ii.) after the end of treatment (month 6) and iii.) at 12 and 18 months follow-up. A tissue sample will also be taken at the time of diagnosis. The blood samples will be used to investigate whether immunological biomarkers such as HSP90, IL1b, IL6, IL10, IL-17, IL1βRa, IL1-RII, HPX, CFB, APOA4 and Serpin-F1-can provide prognostic information related to the development of fatigue in breast cancer patients.

   DNA methylation will be examined by Full-genome methylation assays using Illumina's Human Methylation 850K platform and 8 CpG sites from our partner Mylin Torres will in addition be validated.
9. Data flow

   The REBECCA system will function as a data collection system, and will be a "stand alone" system that will have no communication with other systems in the hospital.

   i.) A smartwatch: The smartwatch to be used in REBECCA for RWD collection will be a commercial Garmin-type smartwatch.

   ii.) REBECCAs patient app (pApp): GPS data, data from third-party health apps, images and sensor data will first be uploaded to REBECCA's pApp. The data will be stored in the app on a separate memory location on the phone, which is isolated and therefore not available for the other phone apps. .

   iii.) REBECCAs PC plug-in: patients will install this on their PC. They will be given a description of how to do this. The connection between the patient ID and REBECCA's browser plug-in will also take place here via a unique code, generated in the pApp on the mobile, which the patient enters into the browser. The user ID is stored so that the patient does not have to log in every time they reopen the browser. The REBECCA's PC plug-in utilizes the browser's local storage space to store information that is critical to its functionality, while the data from the patient's online activity is directly transferred and stored on the REBECCA server for subsequent processing.

   iv.) REBECCAs companion app (cApp): Family members or close friends who will contribute information to REBECCA will report this data in REBECCA's companion app, which they will install on their mobile. .

   v.) RedCap server at HelseVest IKT: Deidentified clinical data and PROM data will be stored in the RedCap server at HelseVest IKT before being transferred pseudonymously and encrypted to the remotely managed REBECCA server.
10. Data storage, privacy and data security

    Data security and privacy are a high priority in REBECCA and will of course be in line with both Norwegian and European laws. The law firm TimeLex, located in Belgium, is responsible for creating an operational data security and ethical framework that the study will follow. This means that all precautions will be taken in REBECCA to respect the privacy of study participants in accordance with European Parliament and Council Regulation (EU) 2016/679 of 27 April 2016 regarding the protection of individuals with regard to the processing of personal data and the free movement of such data , and repealing Directive 95/46 / EC (General Data Protection Regulation) (GDPR))50. TimeLex, will identify and describe the ethical guidelines that apply to the various REBECCA participating countries, and the list of necessary measures will apply to the entire ethical operation of the REBECCA project.
11. Expected impact of the REBECCA project

REBECCA aims to use "real-world data" combined with an advanced data management platform and innovative methods for modeling causal data, to close the gap between clinical research and clinical practice in the treatment of cancer patients. The REBECCA project will initially focus on breast cancer, but will also demonstrate the REBECCA system's transmission to other cancers such as prostate cancer. REBECCA's technological and methodological advances will also be relevant for other clinical research domains that want to investigate the causal relationship between several clinical factors (lifestyle and environmental factors, and comorbidities), through analysis of registry and biobank data and observational data from patients' real life / everyday life.

12 Among REBECCAs milestones are:

A. Development of new approaches to measurement, and a better understanding, of indicators related to the patient's health status and quality of life.

B. Development of methods for statistical and causal analysis of "real-world data".

C. Clinical studies in cancer-related fatigue / fagitue, cancer-induced peripheral neuropathy and cancer-related osteoporosis.

D. Examination of patient monitoring in clinical trials, as a tool to improve the quality of life of cancer patients.

E. Generation and reuse of data sets that will enable the investigation of new medical issues as well as the design, implementation and delivery of an AI-enhanced data collection and management system for comprehensive monitoring of breast cancer survivors' health status and quality of life.

F. To offer new tools and data to clinicians that lead to improved follow-up of cancer patients.

G. Improved patient experience and quality of life due to detailed monitoring and a more personal follow-up.

Digital health (eHealth) has come more into focus during the COVID-19 pandemic. The REBECCA system will be able to contribute to development, increased use and increased competence in eHealth at Stavanger University Hospital by offering digital data collection, digital solutions for patient monitoring, digital solutions for early detection of comorbidities, use of artificial intelligence models as analysis tools, better utilization of health data from health registers and research biobanks as well as offering health care in new ways etc.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients with histologically detectable M0 breast cancer (stage 0-III) who require neoadjuvant or adjuvant endocrine, chemo and / or radiation therapy at least and no more than 3 months before initiation of study.
* Female breast cancer patients between 19 and 80 years of age.
* Patients who have increased their life expectancy beyond the first 3 months after starting treatment.
* Patients who have the ability to understand the protocol and can participate in the follow-up plan.
* Patients who have an absence of psychological, familial, sociological or geographical condition that potentially impedes compliance with the study protocol and follow-up plan.

Exclusion criteria:

* Male breast cancer patients.
* Patients who do not agree to the study protocol.
* Patients with a previous cancer diagnosis (excluding skin cancer treated only by surgery).
* Patients who have previously been treated with some form of chemotherapy / radiation therapy.

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer affects women in 99% of all cases
Study Population: All breast cancer patients who have undergone surgery at SUS, and who meet the inclusion criteria, will be informed about the REBECCA-1 sub-study and written electronic consent will be obtained from those who wish to participate. All potential participants will be women due to the nature of breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Level of fatigue at diagnosis - baseline | This will be done at diagnosis, before treatment.
  Visual Analogue Scale (fVAS), which is a score from 0 to 100 mm marked on a 100 mm line on a paper.
Change from baseline fVAS after treatment 6 months | 6 months after diagnosis and treatment
  fVAS (score from 0 to 100 mm marked on a 100 mm line on paper)
fVAS follow up 12 months | 12 months after diagnosis and treatment
  fVAS (score from 0 to 100 mm marked on a 100 mm line on paper)
fVAS follow up 18 months | 18 months after diagnosis and treatment
  fVAS (score from 0 to 100 mm marked on a 100 mm line on paper)

SECONDARY OUTCOMES:
Activity and sleep disorder measured with a smart watch. | This will be measured at month 6
  We may measure number of steps each day, papttern of movement and sleep quality
Activity and sleep disorder measured with a smart watch. | This will be measured at month 12
  We may measure number of steps each day, papttern of movement and sleep quality
Activity and sleep disorder measured with a smart watch. | This will be measured at month 18
  We may measure number of steps each day, papttern of movement and sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Svein Skeie, PhD, Study Director — Helse Stavanger HF
Locations (1):
- Helse Stavanger HF, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khozin S, Blumenthal GM, Pazdur R. Real-world Data for Clinical Evidence Generation in Oncology. J Natl Cancer Inst. 2017 Nov 1;109(11). doi: 10.1093/jnci/djx187. PMID 29059439
- [Background] Eichler HG, Pignatti F, Schwarzer-Daum B, Hidalgo-Simon A, Eichler I, Arlett P, Humphreys A, Vamvakas S, Brun N, Rasi G. Randomized Controlled Trials Versus Real World Evidence: Neither Magic Nor Myth. Clin Pharmacol Ther. 2021 May;109(5):1212-1218. doi: 10.1002/cpt.2083. Epub 2020 Nov 12. PMID 33063841
- [Background] Hjermstad MJ, Fayers PM, Bjordal K, Kaasa S. Health-related quality of life in the general Norwegian population assessed by the European Organization for Research and Treatment of Cancer Core Quality-of-Life Questionnaire: the QLQ=C30 (+ 3). J Clin Oncol. 1998 Mar;16(3):1188-96. doi: 10.1200/JCO.1998.16.3.1188. PMID 9508207
- [Background] Chalder T, Berelowitz G, Pawlikowska T, Watts L, Wessely S, Wright D, Wallace EP. Development of a fatigue scale. J Psychosom Res. 1993;37(2):147-53. doi: 10.1016/0022-3999(93)90081-p. PMID 8463991
- [Background] Loge JH, Kaasa S. Short form 36 (SF-36) health survey: normative data from the general Norwegian population. Scand J Soc Med. 1998 Dec;26(4):250-8. PMID 9868748
- [Background] Bardsen K, Nilsen MM, Kvaloy JT, Norheim KB, Jonsson G, Omdal R. Heat shock proteins and chronic fatigue in primary Sjogren's syndrome. Innate Immun. 2016 Apr;22(3):162-7. doi: 10.1177/1753425916633236. Epub 2016 Feb 25. PMID 26921255
- [Background] Smith AK, Conneely KN, Pace TW, Mister D, Felger JC, Kilaru V, Akel MJ, Vertino PM, Miller AH, Torres MA. Epigenetic changes associated with inflammation in breast cancer patients treated with chemotherapy. Brain Behav Immun. 2014 May;38:227-36. doi: 10.1016/j.bbi.2014.02.010. Epub 2014 Feb 28. PMID 24583204
- [Background] Curt GA, Breitbart W, Cella D, Groopman JE, Horning SJ, Itri LM, Johnson DH, Miaskowski C, Scherr SL, Portenoy RK, Vogelzang NJ. Impact of cancer-related fatigue on the lives of patients: new findings from the Fatigue Coalition. Oncologist. 2000;5(5):353-60. doi: 10.1634/theoncologist.5-5-353. PMID 11040270
- [Background] Aggarwal BB, Vijayalekshmi RV, Sung B. Targeting inflammatory pathways for prevention and therapy of cancer: short-term friend, long-term foe. Clin Cancer Res. 2009 Jan 15;15(2):425-30. doi: 10.1158/1078-0432.CCR-08-0149. PMID 19147746
- [Background] Bower JE, Ganz PA, Desmond KA, Bernaards C, Rowland JH, Meyerowitz BE, Belin TR. Fatigue in long-term breast carcinoma survivors: a longitudinal investigation. Cancer. 2006 Feb 15;106(4):751-8. doi: 10.1002/cncr.21671. PMID 16400678
- [Background] Andrykowski MA, Curran SL, Lightner R. Off-treatment fatigue in breast cancer survivors: a controlled comparison. J Behav Med. 1998 Feb;21(1):1-18. doi: 10.1023/a:1018700303959. PMID 9547419
- [Background] Lawrence DP, Kupelnick B, Miller K, Devine D, Lau J. Evidence report on the occurrence, assessment, and treatment of fatigue in cancer patients. J Natl Cancer Inst Monogr. 2004;(32):40-50. doi: 10.1093/jncimonographs/lgh027. PMID 15263040
- [Background] Cave A, Kurz X, Arlett P. Real-World Data for Regulatory Decision Making: Challenges and Possible Solutions for Europe. Clin Pharmacol Ther. 2019 Jul;106(1):36-39. doi: 10.1002/cpt.1426. Epub 2019 Apr 10. No abstract available. PMID 30970161
- [Background] Koch L, Jansen L, Herrmann A, Stegmaier C, Holleczek B, Singer S, Brenner H, Arndt V. Quality of life in long-term breast cancer survivors - a 10-year longitudinal population-based study. Acta Oncol. 2013 Aug;52(6):1119-28. doi: 10.3109/0284186X.2013.774461. Epub 2013 Mar 20. PMID 23514583
- [Derived] Stensland M, Bru KF, Austdal M, Dahl IH, Jonsdottir K, Lende TH, Heimvik C, Elve I, Omdal R, van der Giezen M, Kvivik I, Tangeland B, Davidsen L, Hashemi M, Cais A, van Dijk KJ, Seyoum Y, Blafjelldal V, Sola ST, Papadopoulos A, Kiriakidou N, Ioakeimidis I, Diou C, Sarafis I, Delopoulos A, Janssen EAM, Gilje B, Tjensvoll K. Monitoring cancer-related fatigue and quality of life in breast and prostate cancer patients after primary treatment: a study protocol for the REBECCA trials in Norway. Clin Exp Med. 2026 Feb 8;26(1):133. doi: 10.1007/s10238-026-02073-y. PMID 41655181